CLINICAL TRIAL: NCT05126212
Title: Hospi'Senior : Evaluation of the User Experience of an Innovative Hospital Room Prototype Adapted to the Elderly
Brief Title: Evaluation of the User Experience of an Innovative Hospital Room Prototype Adapted to the Elderly
Acronym: HospiSenior-UX
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-127
Record Dates: First submitted 2021-10-06; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: User Experience
Keywords: elderly; hospital room; innovation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients: Patients admitted to the Hospi'Senior room
  Interventions: Other: User experience
- Informal caregivers: Informal caregivers of patients admitted to the Hospi'Senior room
  Interventions: Other: User experience
- Caregivers: Caregivers who have worked in the Hospi'Senior room
  Interventions: Other: User experience

INTERVENTIONS:
Other: User experience — User experience is assessed by validated scale

SUMMARY:
Nowadays in France, the standards of hospital rooms are being questioned in view of the particularities of certain populations admitted to hospitals.

The " Groupement de Coopération Sanitaire des Hôpitaux Universitaires du Grand Ouest " (GCS HUGO) proposes to improve the quality of geriatric care through the modernisation of hospital rooms.

The GCS HUGO has launched a project to co-design a hospital room adapted to the elderly, called "Hospi'Senior", with the help of the "Dependency and Old Age" steering committee. This committee is made up of experts from HUGO and partner companies.

The Hospi'Senior room is composed of innovative technologies concerning bed equipment (e.g. bed canopy), autonomous (e.g. lifeline) and assisted mobility (e.g. rail lift system), lighting (e.g. light guide), communication (touch tablet) and social space (furniture).

The project consists in evaluating the user experience (UX) of :

* patients hospitalized in the Hospi'Senior room,
* informal caregivers of patients hospitalized in the Hospi'Senior room,
* caregivers who have worked in the Hospi'Senior room.

DETAILED DESCRIPTION:
The specificities of Hospi'Senior room are multiple and concern in particular :

* The equipment of the bed :to create a more personalized room: presence of a bed canopy, orientation of the bed towards the windows, presence of a multifunctional space at the head of the bed.
* The autonomous mobility of the patient by facilitating the movements and by preserving the orientation in time of the patient: ephemeris for the temporal orientation, lifeline and sliding door.
* Caregiver-assisted mobility to facilitate patient movements: lifting rail above the bed.
* Lighting to ensure safe movement, especially during the night: light guide, room light, window mirrors, bathroom lighting.
* The digital interface with a touch tablet to improve the occupational and communication aspects.
* The socialization space to welcome visitors in the room.

Design:

Step 1: A visit to the room is made to each participant (patients, informal caregivers, caregivers).

Step 2: no change in care or support for users during hospitalization

Step 3: UX assessment:

* Patients: collected at the end of the hospitalization,
* Informal caregivers: collected at the end of the patient's stay,
* Caregivers: collected after 3 months of using the Hospi'Senior room.

ELIGIBILITY:
Inclusion Criteria:

* Patient :

  * Being admitted to Hospi'Senior room
* Informal caregiver :

  * Be the informal caregiver of a patient admitted to Hospi'Senior room (only one caregiver per patient)
  * Age ≥ 18 years old
  * Able to visit the patient admitted to Hospi'Senior room
* Caregiver :

  * Age ≥ 18 years old
  * Be a healthcare professional involved in the short-term geriatric unit, from one of 4 categories:

    * physicians,
    * permanent paramedical caregivers (nurse, nurse's aide, health executive),
    * support paramedical staff (psychologist, neuropsychologist, physiotherapist, adapted physical activity teacher),
    * technical staff (stretcher bearer).

Exclusion Criteria:

* Patient :

  * Contraindication to participation in the study at the discretion of the medical team
  * Refusal to participate
  * Poor understanding of the French language
  * Persons deprived of liberty by an administrative or judicial decision, persons under forced psychiatric care, adults under legal protection or unable to express their consent
* Informal caregiver :

  * Refusal to participate
  * Poor understanding of the French language
  * Persons deprived of liberty by an administrative or judicial decision, persons under forced psychiatric care, adults under legal protection
* Caregiver :

  * Be a staff in training
  * Less than 3 months seniority in the unit
  * Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Admissions to the Hospi'Senior room are made as the service operates, without prior selection of patients admitted.
  The study is proposed to : i) patients admitted to the Hospi'Senior room, ii) informal caregivers of patients admitted to the Hospi'Senior room, and iii) caregivers who have worked in the Hospi'Senior room.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
User experience of patients (AttrakDiff) | at the end of hospitalization, an average of 9 days
  User experience of the Hospi'Senior room is assessed by Attrakdiff scale (20 items)
User experience of patients (meCUE) | at the end of hospitalization, an average of 9 days
  User experience of the Hospi'Senior room is assessed by meCUE (Modular Evaluation of key Components of User Experience) scale module 2 (8 items)

SECONDARY OUTCOMES:
User experience of informal caregivers (Attrakdiff) | at the end of hospitalization, an average of 9 days
  User experience of the Hospi'Senior room is assessed by Attrakdiff scale (20 items)
User experience of informal caregivers (meCUE) | at the end of hospitalization, an average of 9 days
  User experience of the Hospi'Senior room is assessed by meCUE scale module 2 (8 items)
User experience of caregivers (AttrakDiff) | after 3 months of using the Hospi'Senior room
  User experience of the Hospi'Senior room is assessed by Attrakdiff scale (20 items)
User experience of caregivers (meCUE) | after 3 months of using the Hospi'Senior room
  User experience of the Hospi'Senior room is assessed by meCUE scale module 2 (8 items)
User experience of patients and informal caregivers of each equipment | at the end of hospitalization, an average of 9 days
  User experience of each equipment is assessed by meCUE module 1 (5 items)
User experience of caregivers of each equipment | after 3 months of using the Hospi'Senior room
  User experience of each equipment is assessed by meCUE module 1 (5 items)
Safety aspect of "mobility" and "lighting" equipment | at the end of hospitalization, an average of 9 days
  Safety aspect is assessed by QUEST (Quebec User Evaluation of Satisfaction with assistive Technology) scale for patients and informal caregivers
Safety aspect of "mobility" and "lighting" equipment | after 3 months of using the Hospi'Senior room
  Safety aspect is assessed by QUEST scale for caregivers
Felt affects by caregivers | after 3 months of using the Hospi'Senior room
  Felt affects are assessed by PANAS (Positive And Negative Affect Schedule) scale (20 items)

CONTACTS AND LOCATIONS:
Overall Officials: Cédric ANNWEILER, MD,PhD, Principal Investigator — Angers University Hospital